CLINICAL TRIAL: NCT01324089
Title: A Randomized, Double-Blind Pilot Trial of Resveratrol With or Without Piperine to Enhance Plasma Levels of Resveratrol
Brief Title: Resveratrol With or Without Piperine to Enhance Plasma Levels of Resveratrol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CO 10308; R21CA149560 (NIH); A534260 (Other: UW Madison); SMPH\MEDICINE\HEM-ONC (Other: UW Madison); NCI-2012-00072 (Registry Identifier: NCI Trial ID); 2010-0356 (Other: Institutional Review Board)
Record Dates: First submitted 2011-03-08; First posted 2011-03-28 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2013-05

CONDITIONS: Focus of the Study: Normal Volunteers
Keywords: Resveratrol; Piperine
MeSH Terms: interventions — Resveratrol; piperine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 (Active Comparator): Resveratrol 2.5 grams x 1 dose
  Interventions: Dietary Supplement: Resveratrol
- Arm 2 (Experimental): Resveratrol 2.5 grams x 1 dose and Piperine 5 mg x 1 dose
  Interventions: Dietary Supplement: Resveratrol 2.5 grams x 1 dose and Piperine 5 mg x 1 dose
- Arm 3 (Other): Resveratrol 2.5 grams x 1 dose and Piperine 25 mg x 1 dose
  Interventions: Dietary Supplement: Resveratrol 2.5 grams x 1 dose and Piperine 25 mg x 1 dose

INTERVENTIONS:
Dietary Supplement: Resveratrol — Resveratrol 2.5 grams
  Arms: Arm 1
Dietary Supplement: Resveratrol 2.5 grams x 1 dose and Piperine 5 mg x 1 dose — Resveratrol 2.5 grams x 1 dose and Piperine 5 mg x 1 dose
  Arms: Arm 2
Dietary Supplement: Resveratrol 2.5 grams x 1 dose and Piperine 25 mg x 1 dose — Resveratrol 2.5 grams x 1 dose and Piperine 25 mg x 1 dose
  Arms: Arm 3

SUMMARY:
There is some evidence that when resveratrol (a substance which is found in red grapes, peanuts and chocolate) is combined with Piperine (a substance found in pepper) it is more effective in fighting cancer. The purpose of this study is to see if resveratrol in combination with piperine is more effective than taking resveratrol alone. Since investigators don't know what dose of piperine to use in combination with resveratrol, two different doses of piperine will be studied.

Twenty-four participants, equal numbers of males and females, will receive a single dose of resveratrol (2.5 grams) without piperine, resveratrol (2.5 grams) with piperine (5 mg), or resveratrol (2.5 grams) with piperine (25 mg).

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 18 to 65 years old, inclusive
* Women and men must agree to use an effective form of birth control prior to study entry and for the duration of study participation
* Willingness to abstain from foods containing resveratrol for 3 days prior to single dose administration and for 7 days after dosing. (Examples include red grapes, grape juice, peanuts, peanut butter.)
* Abstain from vitamin supplements from 2 weeks before study dosing and for 7 days following study dosing
* Eastern Cooperative Oncology Group performance status ≤ 1 (Karnofsky > 70%)
* Participants must have normal organ and hepatic functions
* Participants must abstain from alcohol beverages 72 hours prior to dosing with the study agent, and for 7 days after dosing.

Exclusion Criteria:

* Participants who require daily medication, either prescription or over the counter (with the exception of birth control pills) will be considered ineligible. Participants who occasionally use medication (such as for pain relief or allergies) will be considered eligible; however, these participants must agree to refrain from using prn medications starting at midnight prior to the inpatient period and for seven days following dosing.
* Any cancer diagnosis within the past 5 years (except basal cell carcinoma or squamous cell carcinoma).
* Participants may not be currently receiving any other investigational agent(s) or have taken any within the past 9 months.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition of resveratrol and/or piperine.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-03; Primary Completion 2011-11 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Blood levels of study drugs | 30 days
  Blood levels of Resveratrol/Piperine will be measured

SECONDARY OUTCOMES:
Side effects of study drugs | 30 days
  Adverse events or side effects

CONTACTS AND LOCATIONS:
Overall Officials: Howard H Bailey, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States